CLINICAL TRIAL: NCT01559415
Title: An Adipocyte-Driven Mechanism For Weight Regain After Weight Loss: The Yo-Yo Effect
Acronym: ADIPOSTRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 38099
Record Dates: First submitted 2012-03-12; First posted 2012-03-21 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Obesity; Weight Loss; Diet
Keywords: Adipocytes
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Very Low Calorie Diet (Experimental)
  Interventions: Other: Meal replacement diet using Modifast
- Low Calorie Diet (Active Comparator): 1250 kcal diet in which Modifast is given in combination with a normal diet
  Interventions: Other: Normal diet combined with Modifast diet

INTERVENTIONS:
Other: Meal replacement diet using Modifast — modifast intensive diet replacing all regular meals (500 kcal/d) for 5 weeks
  Arms: Very Low Calorie Diet
Other: Normal diet combined with Modifast diet — Combination of modifast and regular diet (1250 kcal/d) for 3 months
  Arms: Low Calorie Diet

SUMMARY:
Almost half of the Dutch population is currently characterized by overweight and obesity. Losing weight is not the problem in obesity treatment, it is the seemingly obligatory weight regain after weight loss: the yoyo-effect. The primary objective of this study is to investigate the association between the weight-loss-induced cellular stress response and the rate of weight regain. The secondary objective is to investigate the differences in cellular stress response and weight regain after rapid and slow weight loss. To investigate this, subjects will receive meal replacements replacing either all or part of the daily meals during the intervention period. THe first group will consume 500 kcal/d diet for 5 weeks while the second group consumes a 1250 kcal/d diet for 3 months, both followed by 1 week normalization and a 2 week strict weight maintenance diet. During the 9-month follow-up period subjects will receive dietary advice according to the Dutch recommendations for healthy eating. The association between the amount of weight regain after the weight loss period and changes in adipokines, parameters of adipocyte metabolism, in vivo adipose tissue metabolism, adipocyte extracellular matrix gene expression profiles, adipocyte stress protein expression and gene polymorphisms in selected genes.

ELIGIBILITY:
Inclusion Criteria:

* Age (years): 20-65
* Body Mass Index (kg/m2): 28-35
* Non-smokers

Exclusion Criteria:

* Subjects using prescription medication, or suffering from diseases or conditions that might influence the outcome of the study: this concerns diseases/medication that influence body weight regulation (malabsorption, untreated hypo/hyperthyroidism, eating disorders, systemic use of steroids, etc.) and obesity-related cardiovascular risk factors (heart disease, systolic and diastolic blood pressures > 160/100 mmHg, blood glucose > 6.1 mmol L-1, blood cholesterol > 7 mmol L-1, blood triglycerides > 3 mmol L-1)
* marked alcohol consumption > 21 alcoholic units week-1 (male), or >14 alcoholic units week-1 (female)
* planned major changes in physical activity during the study to an extent that might interfere with the study outcome as judged by the investigator;
* blood donation within the past 2 months prior to the study
* weight change of >3 kg within 2 months prior to the study
* psychiatric disease (based on medical history only)
* pregnant or lactating women, or women planning to become pregnant within the next 12 months
* surgically treated obesity
* participation in other clinical studies within the last 3 months
* drug abuse (based on clinical judgment)
* unable to give informed consent
* unable to engage in a low-calorie diet
* unable to lose more then 8% of body weight after weight-loss period
* following a special diet (vegetarian, Atkins or other).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
change in weight following weight loss | at 9 weeks and at 46 weeks
  VLCD diet group
change in weight following weight loss | at 16 weeks and at 53 weeks
  LCD diet group

SECONDARY OUTCOMES:
change in adipokine profile due to dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
  In VLCD-group.
  Parameters of adipokine profile, including:
  leptin, acylation stimulating protein (ASP/C3adesarg), adiponectin, resistin, IL-6, RBP4, PAI-1, ACE, FGF-21, Vaspin, Apelin, Nesfatin-1 and TNFa
change in adipokine during weight stable-period (VLCD-group) | after 5 weeks of VLCD diet and after 9 weeks
  In VLCD-group.
  Parameters of adipokine profile, including:
  leptin, acylation stimulating protein (ASP/C3adesarg), adiponectin, resistin, IL-6, RBP4, PAI-1, ACE, FGF-21, Vaspin, Apelin, Nesfatin-1 and TNFa
change in adipokine profile during follow-up (VLCD-group) | at 9 weeks and after follow-up at 46 weeks
  In VLCD-group.
  Parameters of adipokine profile, including:
  leptin, acylation stimulating protein (ASP/C3adesarg), adiponectin, resistin, IL-6, RBP4, PAI-1, ACE, FGF-21, Vaspin, Apelin, Nesfatin-1 and TNFa
change in adipokine profile due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
  In LCD-group.
  Parameters of adipokine profile, including:
  leptin, acylation stimulating protein (ASP/C3adesarg), adiponectin, resistin, IL-6, RBP4, PAI-1, ACE, FGF-21, Vaspin, Apelin, Nesfatin-1 and TNFa
change in adipokine profile during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at 16 weeks
  In LCD-group.
  Parameters of adipokine profile, including:
  leptin, acylation stimulating protein (ASP/C3adesarg), adiponectin, resistin, IL-6, RBP4, PAI-1, ACE, FGF-21, Vaspin, Apelin, Nesfatin-1 and TNFa
change in adipokine profile during follow-up (LCD-group) | at 16 weeks and after follow-up at 53 weeks
  In LCD-group.
  Parameters of adipokine profile, including:
  leptin, acylation stimulating protein (ASP/C3adesarg), adiponectin, resistin, IL-6, RBP4, PAI-1, ACE, FGF-21, Vaspin, Apelin, Nesfatin-1 and TNFa
Changes in adipokine profile in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In LCD-group.
  Parameters of adipokine profile, including:
  leptin, acylation stimulating protein (ASP/C3adesarg), adiponectin, resistin, IL-6, RBP4, PAI-1, ACE, FGF-21, Vaspin, Apelin, Nesfatin-1 and TNFa
change in adipokine profile in relation to weight regain during follow-up | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In LCD-group and VLCD-group
  Parameters of adipokine profile, including:
  leptin, acylation stimulating protein (ASP/C3adesarg), adiponectin, resistin, IL-6, RBP4, PAI-1, ACE, FGF-21, Vaspin, Apelin, Nesfatin-1 and TNFa
change in parameters of adipocyte fat metabolism due to dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
  In VLCD-group.
  Parameters of adipocyte fat metabolism:
  * ALDOC, phospho-annexin2, FABP4, PLIN-B, HADH, phosphorylated HSL and non-phosphorylated HSL - immunohistochemical staining of GLUT-4
  * Micro-array analysis of gene expression profile
change in parameters of adipocyte fat metabolism during weight-stable period (VLCD-group) | after 5 weeks of VLCD diet and at 9 weeks
  In VLCD-group.
  Parameters of adipocyte fat metabolism:
  * ALDOC, phospho-annexin2, FABP4, PLIN-B, HADH, phosphorylated HSL and non-phosphorylated HSL - immunohistochemical staining of GLUT-4
  * Micro-array analysis of gene expression profile
change in parameters of adipocyte fat metabolism during follow-up period (VLCD-group) | at 9 weeks and after follow-up at 46 weeks
  In VLCD-group.
  Parameters of adipocyte fat metabolism:
  * ALDOC, phospho-annexin2, FABP4, PLIN-B, HADH, phosphorylated HSL and non-phosphorylated HSL - immunohistochemical staining of GLUT-4
  * Micro-array analysis of gene expression profile
change in parameters of adipocyte fat metabolism due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
  In LCD-group.
  Parameters of adipocyte fat metabolism:
  * ALDOC, phospho-annexin2, FABP4, PLIN-B, HADH, phosphorylated HSL and non-phosphorylated HSL - immunohistochemical staining of GLUT-4
  * Micro-array analysis of gene expression profile
change in parameters of adipocyte fat metabolism during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at 16 weeks
  In LCD-group.
  Parameters of adipocyte fat metabolism:
  * ALDOC, phospho-annexin2, FABP4, PLIN-B, HADH, phosphorylated HSL and non-phosphorylated HSL - immunohistochemical staining of GLUT-4
  * Micro-array analysis of gene expression profile
change in parameters of adipocyte fat metabolism during follow-up (LCD-group) | at 16 weeks and after follow-up at 53 weeks
  In LCD-group.
  Parameters of adipocyte fat metabolism:
  * ALDOC, phospho-annexin2, FABP4, PLIN-B, HADH, phosphorylated HSL and non-phosphorylated HSL - immunohistochemical staining of GLUT-4
  * Micro-array analysis of gene expression profile
Changes in parameters of adipocyte fat metabolism in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  Parameters of adipocyte fat metabolism:
  * ALDOC, phospho-annexin2, FABP4, PLIN-B, HADH, phosphorylated HSL and non-phosphorylated HSL - immunohistochemical staining of GLUT-4
  * Micro-array analysis of gene expression profile
change in parameters of adipocyte fat metabolism in relation to weight regain during follow-up | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In LCD-group and VLCD-group.
  Parameters of adipocyte fat metabolism:
  * ALDOC, phospho-annexin2, FABP4, PLIN-B, HADH, phosphorylated HSL and non-phosphorylated HSL - immunohistochemical staining of GLUT-4
  * Micro-array analysis of gene expression profile
change in in-vivo adipose tissue metabolism due to dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
  In VLCD-group.
  In-vivo adipose tissue metabolism assessed in fasting and postprandial conditions:
  * adipose tissue blood flow
  * adipose tissue PO2
  * adipose tissue oxygen consumption
  * adipose tissue capacity for fat uptake from chylomicron-triglycerides
change in in-vivo adipose tissue metabolism during weight-stable period (VLCD-group) | after 5 weeks of VLCD diet and at 9 weeks
  In VLCD-group.
  In-vivo adipose tissue metabolism assessed in fasting and postprandial conditions:
  * adipose tissue blood flow
  * adipose tissue PO2
  * adipose tissue oxygen consumption
  * adipose tissue capacity for fat uptake from chylomicron-triglycerides
change in in-vivo adipose tissue metabolism during follow-up period (VLCD-group) | at 9 weeks and after follow-up period at 46 weeks
  In VLCD-group.
  In-vivo adipose tissue metabolism assessed in fasting and postprandial conditions:
  * adipose tissue blood flow
  * adipose tissue PO2
  * adipose tissue oxygen consumption
  * adipose tissue capacity for fat uptake from chylomicron-triglycerides
change in in-vivo adipose tissue metabolism due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
  In LCD-group.
  In-vivo adipose tissue metabolism assessed in fasting and postprandial conditions:
  * adipose tissue blood flow
  * adipose tissue PO2
  * adipose tissue oxygen consumption
  * adipose tissue capacity for fat uptake from chylomicron-triglycerides
change in in-vivo adipose tissue metabolism during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at 16 weeks
  In LCD-group.
  In-vivo adipose tissue metabolism assessed in fasting and postprandial conditions:
  * adipose tissue blood flow
  * adipose tissue PO2
  * adipose tissue oxygen consumption
  * adipose tissue capacity for fat uptake from chylomicron-triglycerides
change in in-vivo adipose tissue metabolism during follow-up period (LCD-group) | at 16 weeks and after follow-up period at 53 weeks
  In LCD-group.
  In-vivo adipose tissue metabolism assessed in fasting and postprandial conditions:
  * adipose tissue blood flow
  * adipose tissue PO2
  * adipose tissue oxygen consumption
  * adipose tissue capacity for fat uptake from chylomicron-triglycerides
change in in-vivo adipose tissue metabolism in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In-vivo adipose tissue metabolism assessed in fasting and postprandial conditions:
  * adipose tissue blood flow
  * adipose tissue PO2
  * adipose tissue oxygen consumption
  * adipose tissue capacity for fat uptake from chylomicron-triglycerides
change in in-vivo adipose tissue metabolism in relation to weight regain during follow-up | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In LCD-group and VLCD-group
  In-vivo adipose tissue metabolism assessed in fasting and postprandial conditions:
  * adipose tissue blood flow
  * adipose tissue PO2
  * adipose tissue oxygen consumption
  * adipose tissue capacity for fat uptake from chylomicron-triglycerides
change in the adipocyte extracellular matrix gene and protein expression profile due to dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
  VLCD diet group
  Adipocyte extracellular matrix gene expression profile assessed:
  * micro-arrays on RNA expression
  * protein expression
  * Genetic polymorphisms: focus on polymorphisms in genes (a) that are preferentially expressed in white adipose tissue like TIMP4, (b) that have a proposed anchoring role of the cells to the basal lamina like the non-fibrillar type collagens IV and VI, (c) that are essential for adipose tissue development like MMP14, and (d) for which association has been found with obesity or adiposity like TIMP1, MMP2 and MMP9
change in the adipocyte extracellular matrix gene and protein expression profile during weight-stable period (VLCD-group) | after 5 weeks of VLCD diet and at 9 weeks
  VLCD diet group
  Adipocyte extracellular matrix gene expression profile assessed:
  * micro-arrays on RNA expression
  * protein expression
  * Genetic polymorphisms: focus on polymorphisms in genes (a) that are preferentially expressed in white adipose tissue like TIMP4, (b) that have a proposed anchoring role of the cells to the basal lamina like the non-fibrillar type collagens IV and VI, (c) that are essential for adipose tissue development like MMP14, and (d) for which association has been found with obesity or adiposity like TIMP1, MMP2 and MMP9
change in the adipocyte extracellular matrix gene and protein expression profile during follow-up period (VLCD-group) | at 9 weeks and after follow-up period at 46 weeks
  VLCD diet group
  Adipocyte extracellular matrix gene expression profile assessed:
  * micro-arrays on RNA expression
  * protein expression
  * Genetic polymorphisms: focus on polymorphisms in genes (a) that are preferentially expressed in white adipose tissue like TIMP4, (b) that have a proposed anchoring role of the cells to the basal lamina like the non-fibrillar type collagens IV and VI, (c) that are essential for adipose tissue development like MMP14, and (d) for which association has been found with obesity or adiposity like TIMP1, MMP2 and MMP9
change in the adipocyte extracellular matrix gene and protein expression profile due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
  LCD diet group
  Adipocyte extracellular matrix gene expression profile assessed:
  * micro-arrays on RNA expression
  * protein expression
  * Genetic polymorphisms: focus on polymorphisms in genes (a) that are preferentially expressed in white adipose tissue like TIMP4, (b) that have a proposed anchoring role of the cells to the basal lamina like the non-fibrillar type collagens IV and VI, (c) that are essential for adipose tissue development like MMP14, and (d) for which association has been found with obesity or adiposity like TIMP1, MMP2 and MMP9
change in the adipocyte extracellular matrix gene and protein expression profile during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at 16 weeks
  LCD diet group
  Adipocyte extracellular matrix gene expression profile assessed:
  * micro-arrays on RNA expression
  * protein expression
  * Genetic polymorphisms: focus on polymorphisms in genes (a) that are preferentially expressed in white adipose tissue like TIMP4, (b) that have a proposed anchoring role of the cells to the basal lamina like the non-fibrillar type collagens IV and VI, (c) that are essential for adipose tissue development like MMP14, and (d) for which association has been found with obesity or adiposity like TIMP1, MMP2 and MMP9
change in the adipocyte extracellular matrix gene and protein expression profile during follow-up period (LCD-group) | at 16 weeks and after follow-up period
  LCD diet group
  Adipocyte extracellular matrix gene expression profile assessed:
  * micro-arrays on RNA expression
  * protein expression
  * Genetic polymorphisms: focus on polymorphisms in genes (a) that are preferentially expressed in white adipose tissue like TIMP4, (b) that have a proposed anchoring role of the cells to the basal lamina like the non-fibrillar type collagens IV and VI, (c) that are essential for adipose tissue development like MMP14, and (d) for which association has been found with obesity or adiposity like TIMP1, MMP2 and MMP9
change in the adipocyte extracellular matrix gene and protein expression profile in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  Adipocyte extracellular matrix gene expression profile assessed:
  * micro-arrays on RNA expression
  * protein expression
  * Genetic polymorphisms: focus on polymorphisms in genes (a) that are preferentially expressed in white adipose tissue like TIMP4, (b) that have a proposed anchoring role of the cells to the basal lamina like the non-fibrillar type collagens IV and VI, (c) that are essential for adipose tissue development like MMP14, and (d) for which association has been found with obesity or adiposity like TIMP1, MMP2 and MMP9
change in the adipocyte extracellular matrix gene and protein expression profile in relation to weight regain during follow-up | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In LCD-group and VLCD-group
  Adipocyte extracellular matrix gene expression profile assessed:
  * micro-arrays on RNA expression
  * protein expression
  * Genetic polymorphisms: focus on polymorphisms in genes (a) that are preferentially expressed in white adipose tissue like TIMP4, (b) that have a proposed anchoring role of the cells to the basal lamina like the non-fibrillar type collagens IV and VI, (c) that are essential for adipose tissue development like MMP14, and (d) for which association has been found with obesity or adiposity like TIMP1, MMP2 and MMP9
change in adipocyte stress proteins expression due to dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
  VLCD diet group
  Adipocyte stress proteins expression:
  * components of stress fibers and focal adhesions, like integrins
  * 43 'stress proteins' with focus on 9 stress proteins: actin betaactin, gamma 1, Rho GDP dissociation inhibitor (GDI), alphacofilin 1 (non-muscle), keratin 8, stathmin 1/oncoprotein 18, tropomyosin 3, vimentin, tubulin beta
change in adipocyte stress proteins expression during weight-stable period (VLCD-group) | after 5 weeks of VLCD diet and at 9 weeks
  VLCD diet group
  Adipocyte stress proteins expression:
  * components of stress fibers and focal adhesions, like integrins
  * 43 'stress proteins' with focus on 9 stress proteins: actin betaactin, gamma 1, Rho GDP dissociation inhibitor (GDI), alphacofilin 1 (non-muscle), keratin 8, stathmin 1/oncoprotein 18, tropomyosin 3, vimentin, tubulin beta
change in adipocyte stress proteins expression during follow-up period (VLCD-group) | at 9 weeks and after follow-up period at week 46
  VLCD diet group
  Adipocyte stress proteins expression:
  * components of stress fibers and focal adhesions, like integrins
  * 43 'stress proteins' with focus on 9 stress proteins: actin betaactin, gamma 1, Rho GDP dissociation inhibitor (GDI), alphacofilin 1 (non-muscle), keratin 8, stathmin 1/oncoprotein 18, tropomyosin 3, vimentin, tubulin beta
change in adipocyte stress proteins expression due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
  LCD diet group
  Adipocyte stress proteins expression:
  * components of stress fibers and focal adhesions, like integrins
  * 43 'stress proteins' with focus on 9 stress proteins: actin betaactin, gamma 1, Rho GDP dissociation inhibitor (GDI), alphacofilin 1 (non-muscle), keratin 8, stathmin 1/oncoprotein 18, tropomyosin 3, vimentin, tubulin beta
change in adipocyte stress proteins expression during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at week 16
  LCD diet group
  Adipocyte stress proteins expression:
  * components of stress fibers and focal adhesions, like integrins
  * 43 'stress proteins' with focus on 9 stress proteins: actin betaactin, gamma 1, Rho GDP dissociation inhibitor (GDI), alphacofilin 1 (non-muscle), keratin 8, stathmin 1/oncoprotein 18, tropomyosin 3, vimentin, tubulin beta
change in adipocyte stress proteins expression during follow-up period (LCD-group) | at week 16 and after follow-up period at 53 weeks
  LCD diet group
  Adipocyte stress proteins expression:
  * components of stress fibers and focal adhesions, like integrins
  * 43 'stress proteins' with focus on 9 stress proteins: actin betaactin, gamma 1, Rho GDP dissociation inhibitor (GDI), alphacofilin 1 (non-muscle), keratin 8, stathmin 1/oncoprotein 18, tropomyosin 3, vimentin, tubulin beta
change in adipocyte stress proteins expression in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  Adipocyte stress proteins expression:
  * components of stress fibers and focal adhesions, like integrins
  * 43 'stress proteins' with focus on 9 stress proteins: actin betaactin, gamma 1, Rho GDP dissociation inhibitor (GDI), alphacofilin 1 (non-muscle), keratin 8, stathmin 1/oncoprotein 18, tropomyosin 3, vimentin, tubulin beta
change in adipocyte stress proteins expression in relation to weight regain during follow-up | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In LCD-group and VLCD-group
  Adipocyte stress proteins expression:
  * components of stress fibers and focal adhesions, like integrins
  * 43 'stress proteins' with focus on 9 stress proteins: actin betaactin, gamma 1, Rho GDP dissociation inhibitor (GDI), alphacofilin 1 (non-muscle), keratin 8, stathmin 1/oncoprotein 18, tropomyosin 3, vimentin, tubulin beta
change in physiological parameters due to dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
  Physiological parameters:
  Blood pressure, waist-, and hip-circumference, weight, BMI, age, body fat
change in physiological parameters during weight-stable period (VLCD-group) | after 5 weeks of VLCD diet and at 9 weeks
  Physiological parameters:
  Blood pressure, waist-, and hip-circumference, weight, BMI, age, body fat
change in physiological parameters during follow-up period (VLCD-group) | at 9 weeks and after follow-up at 46 weeks
  Physiological parameters:
  Blood pressure, waist-, and hip-circumference, weight, BMI, age, body fat
change in physiological parameters due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
  Physiological parameters:
  Blood pressure, waist-, and hip-circumference, weight, BMI, age, body fat
change in physiological parameters during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at 16 weeks
  Physiological parameters:
  Blood pressure, waist-, and hip-circumference, weight, BMI, age, body fat
change in physiological parameters during follow-up (LCD-group) | at 16 weeks and after follow-up at 53 weeks
  Physiological parameters:
  Blood pressure, waist-, and hip-circumference, weight, BMI, age, body fat
Changes in physiological parameters in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  Physiological parameters:
  Blood pressure, waist-, and hip-circumference, weight, BMI, age, body fat
Changes in physiological parameters in relation to weight regain during follow-up | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  Physiological parameters:
  Blood pressure, waist-, and hip-circumference, weight, BMI, age, body fat
change in plasma metabolic parameters due to dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
  Plasma metabolic parameters are measured in fasting and postprandial conditions, focused on:
  Glucose, insulin, free fatty acid, glycerol and triglycerides
change in plasma metabolic parameters during weight-stable period (VLCD-group) | after 5 weeks of VLCD diet and at 9 weeks
  Plasma metabolic parameters are measured in fasting and postprandial conditions, focused on:
  Glucose, insulin, free fatty acid, glycerol and triglycerides
change in plasma metabolic parameters during follow-up period (VLCD-group) | at 9 weeks and after follow-up at 46 weeks
  Plasma metabolic parameters are measured in fasting and postprandial conditions, focused on:
  Glucose, insulin, free fatty acid, glycerol and triglycerides
change in plasma metabolic parameters due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
  Plasma metabolic parameters are measured in fasting and postprandial conditions, focused on:
  Glucose, insulin, free fatty acid, glycerol and triglycerides
change in plasma metabolic parameters during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at 16 weeks
  Plasma metabolic parameters are measured in fasting and postprandial conditions, focused on:
  Glucose, insulin, free fatty acid, glycerol and triglycerides
change in plasma metabolic parameters during follow-up (LCD-group) | at 16 weeks and after follow-up at 53 weeks
  Plasma metabolic parameters are measured in fasting and postprandial conditions, focused on:
  Glucose, insulin, free fatty acid, glycerol and triglycerides
Changes in plasma metabolic parameters in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  Plasma metabolic parameters are measured in fasting and postprandial conditions, focused on:
  Glucose, insulin, free fatty acid, glycerol and triglycerides
Changes in plasma metabolic parameters in relation to weight regain during follow-up | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In LCD-group and VLCD-group
  Plasma metabolic parameters are measured in fasting and postprandial conditions, focused on:
  Glucose, insulin, free fatty acid, glycerol and triglycerides
change in fat cell size and fat cell number due to the dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
change in fat cell size and fat cell number during weight-stable period (VLCD-group) | after 5 weeks of VLCD diet and at 9 weeks
change in fat cell size and fat cell number during follow-up period (VLCD-group) | at 9 weeks and after follow-up at 46 weeks
change in fat cell size and fat cell number due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
change in fat cell size and fat cell number during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at 16 weeks
change in fat cell size and fat cell number during follow-up (LCD-group) | at 16 weeks and after follow-up at 53 weeks
Changes in fat cell size and fat cell number in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
Changes in fat cell size and fat cell number in relation to weight regain after weight loss | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In LCD-group and VLCD-group
change in breath volatile organic compounds due to the dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
change in breath volatile organic compounds during weight-stable period (VLCD-group) | after 5 weeks of VLCD diet and at 9 weeks
change in breath volatile organic compounds during follow-up period (VLCD-group) | at 9 weeks and after follow-up at 46 weeks
change in breath volatile organic compounds due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
change in breath volatile organic compounds during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at 16 weeks
change in breath volatile organic compounds during follow-up (LCD-group) | at 16 weeks and after follow-up at 53 weeks
Changes in breath volatile organic compounds in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
Changes in breath volatile organic compounds in relation to weight regain during follow-up | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In LCD-group and VLCD-group
change in inflammatory parameters due to the dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
  In VLCD-group.
  Inflammatory parameters are analyzed in:
  * Plasma (including: TNF-a, IL-6, IL-8 and MCP-1)
  * Micro-array
  * PCR: (including: TNF-a, IL-6, IL-8 and MCP-1)
change in inflammatory parameters during weight-stable period (VLCD-group) | after 5 weeks of VLCD diet and at 9 weeks
  In VLCD-group.
  Inflammatory parameters are analyzed in:
  * Plasma (including: TNF-a, IL-6, IL-8 and MCP-1)
  * Micro-array
  * PCR: (including: TNF-a, IL-6, IL-8 and MCP-1)
change in inflammatory parameters during follow-up period (VLCD-group) | at 9 weeks and after follow-up at 46 weeks
  In VLCD-group.
  Inflammatory parameters are analyzed in:
  * Plasma (including: TNF-a, IL-6, IL-8 and MCP-1)
  * Micro-array
  * PCR: (including: TNF-a, IL-6, IL-8 and MCP-1)
change in inflammatory parameters due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
  In LCD-group.
  Inflammatory parameters are analyzed in:
  * Plasma (including: TNF-a, IL-6, IL-8 and MCP-1)
  * Micro-array
  * PCR: (including: TNF-a, IL-6, IL-8 and MCP-1)
change in inflammatory parameters during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at 16 weeks
  In LCD-group.
  Inflammatory parameters are analyzed in:
  * Plasma (including: TNF-a, IL-6, IL-8 and MCP-1)
  * Micro-array
  * PCR: (including: TNF-a, IL-6, IL-8 and MCP-1)
change in inflammatory parameters during follow-up (LCD-group) | at 16 weeks and after follow-up at 53 weeks
  In LCD-group.
  Inflammatory parameters are analyzed in:
  * Plasma (including: TNF-a, IL-6, IL-8 and MCP-1)
  * Micro-array
  * PCR: (including: TNF-a, IL-6, IL-8 and MCP-1)
Changes in inflammatory parameters in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  Inflammatory parameters are analyzed in:
  * Plasma (including: TNF-a, IL-6, IL-8 and MCP-1)
  * Micro-array
  * PCR: (including: TNF-a, IL-6, IL-8 and MCP-1)
Changes in inflammatory parameters in relation to weight regain during the follow-up | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  Inflammatory parameters are analyzed in:
  * Plasma (including: TNF-a, IL-6, IL-8 and MCP-1)
  * Micro-array
  * PCR: (including: TNF-a, IL-6, IL-8 and MCP-1)
Changes in protein concentration of metabolic parameters due to the dietary intervention (VLCD-group) | at baseline and after 5 weeks of VLCD diet
  Protein concentrations of metabolic parameters, including:
  CD36, FABP4, Vimentin, Vimentin25, HSL, ALDOC, ALDOA, TUBB5, ANXA2, HADH, ACAA2 and ACADS
Changes in protein concentration of metabolic parameters during weight-stable period (VLCD-group) | after 5 weeks of VLCD diet and at 9 weeks
  Protein concentrations of metabolic parameters, including:
  CD36, FABP4, Vimentin, Vimentin25, HSL, ALDOC, ALDOA, TUBB5, ANXA2, HADH, ACAA2 and ACADS
change in protein concentration of metabolic parameters during follow-up (VLCD-group) | at 9 weeks and after follow-up at 46 weeks
  Protein concentrations of metabolic parameters, including:
  CD36, FABP4, Vimentin, Vimentin25, HSL, ALDOC, ALDOA, TUBB5, ANXA2, HADH, ACAA2 and ACADS
change in protein concentration of metabolic parameters due to dietary intervention (LCD-group) | at baseline and after 12 weeks of LCD diet
  Protein concentrations of metabolic parameters, including:
  CD36, FABP4, Vimentin, Vimentin25, HSL, ALDOC, ALDOA, TUBB5, ANXA2, HADH, ACAA2 and ACADS
change in protein concentration of metabolic parameters during weight-stable period (LCD-group) | after 12 weeks of LCD diet and at 16 weeks
  Protein concentrations of metabolic parameters, including:
  CD36, FABP4, Vimentin, Vimentin25, HSL, ALDOC, ALDOA, TUBB5, ANXA2, HADH, ACAA2 and ACADS
change in protein concentration of metabolic parameters during follow-up (LCD-group) | at 16 weeks and after follow-up at 53 weeks
  Protein concentrations of metabolic parameters, including:
  CD36, FABP4, Vimentin, Vimentin25, HSL, ALDOC, ALDOA, TUBB5, ANXA2, HADH, ACAA2 and ACADS
change in protein concentration of metabolic parameters in the LCD-group compared to the VLCD-group | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  Protein concentrations of metabolic parameters, including:
  CD36, FABP4, Vimentin, Vimentin25, HSL, ALDOC, ALDOA, TUBB5, ANXA2, HADH, ACAA2 and ACADS
change in protein concentration of metabolic parameters in relation to weight regain during follow-up | at baseline, at 5, 9, 12, 16, 46 and 53 weeks
  In LCD-group and VLCD-group
  Protein concentrations of metabolic parameters, including:
  CD36, FABP4, Vimentin, Vimentin25, HSL, ALDOC, ALDOA, TUBB5, ANXA2, HADH, ACAA2 and ACADS

CONTACTS AND LOCATIONS:
Overall Officials: Marleen van Baak, Professor, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Qiao Q, Bouwman FG, van Baak MA, Roumans NJT, Vink RG, Mariman ECM. Plasma Levels of Triglycerides and IL-6 Are Associated With Weight Regain and Fat Mass Expansion. J Clin Endocrinol Metab. 2022 Jun 16;107(7):1920-1929. doi: 10.1210/clinem/dgac198. PMID 35366329
- [Derived] Tareen SHK, Kutmon M, de Kok TM, Mariman ECM, van Baak MA, Evelo CT, Adriaens ME, Arts ICW. Stratifying cellular metabolism during weight loss: an interplay of metabolism, metabolic flexibility and inflammation. Sci Rep. 2020 Feb 3;10(1):1651. doi: 10.1038/s41598-020-58358-z. PMID 32015415
- [Derived] Roumans NJT, Wang P, Vink RG, van Baak MA, Mariman ECM. Combined Analysis of Stress- and ECM-Related Genes in Their Effect on Weight Regain. Obesity (Silver Spring). 2018 Mar;26(3):492-498. doi: 10.1002/oby.22093. Epub 2018 Feb 5. PMID 29399976
- [Derived] Vink RG, Roumans NJ, van der Kolk BW, Fazelzadeh P, Boekschoten MV, Mariman EC, van Baak MA. Adipose Tissue Meal-Derived Fatty Acid Uptake Before and After Diet-Induced Weight Loss in Adults with Overweight and Obesity. Obesity (Silver Spring). 2017 Aug;25(8):1391-1399. doi: 10.1002/oby.21903. Epub 2017 Jun 22. PMID 28639346
- [Derived] Roumans NJ, Vink RG, Fazelzadeh P, van Baak MA, Mariman EC. A role for leukocyte integrins and extracellular matrix remodeling of adipose tissue in the risk of weight regain after weight loss. Am J Clin Nutr. 2017 May;105(5):1054-1062. doi: 10.3945/ajcn.116.148874. Epub 2017 Mar 15. PMID 28298393
- [Derived] Vink RG, Roumans NJ, Cajlakovic M, Cleutjens JPM, Boekschoten MV, Fazelzadeh P, Vogel MAA, Blaak EE, Mariman EC, van Baak MA, Goossens GH. Diet-induced weight loss decreases adipose tissue oxygen tension with parallel changes in adipose tissue phenotype and insulin sensitivity in overweight humans. Int J Obes (Lond). 2017 May;41(5):722-728. doi: 10.1038/ijo.2017.38. Epub 2017 Feb 9. PMID 28179648